CLINICAL TRIAL: NCT06690281
Title: A Phase II Study of Adjuvant Immunotherapy Targeting KRAS G12D, KRAS G12V, or TP53 R175H for Participants With Advanced Gastrointestinal Malignancies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left NIH.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001870; 001870-C
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Carcinoma; Pancreatic Cancer; Hepatocellular Cancer; Cholangiocarcinoma; Duodenal Cancer; Colorectal Cancer; Small Bowel Cancer; Metastatic Cancers
Keywords: KRAS Mutations; Cell Therapy; Gene Therapy; Tp53 Mutations; Immunotherapy; KRAS G12D; KRAS G12V; Tp53; R175H
MeSH Terms: conditions — Pancreatic Neoplasms; Liver Neoplasms; Cholangiocarcinoma; Duodenal Neoplasms; Colorectal Neoplasms; Neoplasms | interventions — aldesleukin; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ TCR T-cells and aldesleukin (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + TCR T cells + aldesleukin
  Interventions: Biological: KRAS TCR-Transduced PBL; Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide
- 2/ No cellular therapy (No Intervention): Surveillance and follow-up

INTERVENTIONS:
Biological: KRAS TCR-Transduced PBL — Day 0: Cells will be infused intravenously (IV) over 20-30 minutes (2-4 days after the last dose of fludarabine)
  Arms: 1/ TCR T-cells and aldesleukin
Drug: Aldesleukin — Aldesleukin 600,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 3 days (maximum 3 doses)
  Arms: 1/ TCR T-cells and aldesleukin
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg/m^2/day IVPB daily over 30 minutes for 4 days
  Arms: 1/ TCR T-cells and aldesleukin
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 30 mg/kg/day x 2 days IV in 250 mL D5W infused simultaneously with mesna 7.5 mg/kg/day over 1 hour x 2 days
  Arms: 1/ TCR T-cells and aldesleukin

SUMMARY:
Background:

Gastrointestinal (GI) cancer affects the organs (such as the stomach, large and small intestine, pancreas, colon, liver, and biliary system) of the digestive tract. In some participants who have had surgery for GI cancer, blood tests show that the cancer has spread despite being unable to be identified by scans. Certain gene mutations (changes) in GI cancer (such as KRAS or TP53) can be targeted by T cells, a type of immune cell, in individuals with specific HLA types (genes that help proteins in the body know what is self and non-self). Researchers want to see if they can stop GI cancer from returning or spreading in people with these gene mutations and specific HLA types.

Objective:

To test therapy with modified T-cells to prevent or delay the return of GI cancer after standard treatment. T-cells play a role in the body s immune system.

Eligibility:

People aged 18 to 72 years with GI cancer that was treated with standard therapy and is not seen on imaging scans. They must have specific gene mutations and HLA types. They also must have certain clinical or blood tests showing the cancer is spreading (elevating CA19-9 or detectable ctDNA).

Design:

Participants will be divided into 2 groups. Participants nor the study team can choose what Group to participate in; this is done by randomization , like flipping a coin. Participants will have a 1-to-1 chance of being in Group 1 or Group 2.

Group 1 will receive T-cell therapy. Their own T-cells will be collected. In a lab, the cells will be combined with a virus that carries a protein to target cancer cells.

Group 1 participants will stay in the hospital for 3 weeks or more. They will have chemotherapy, and their modified T-cells will be infused through a tube attached to a needle inserted into a vein.

Group 1 participants will visit the clinic every 3 months for 1 year and then every 6 months for 5 years. Then they will have follow-up visits for another 10 years under a different protocol.

Group 2 participants will not receive treatment with T-cells. They will visit the clinic every 3 months for 1 year and then every 6 months for 5 years.

DETAILED DESCRIPTION:
Background:

-Despite definitive surgical resection and (neo)adjuvant chemotherapy, many patients with gastrointestinal carcinomas (GIC) remain at high risk of recurrence and disease-specific mortality. This includes virtually all patients with resected pancreas ductal adenocarcinoma

(PDAC), patients with resected colorectal liver, lung, and/or lymph node metastases (CRLM) with persistently elevated circulating tumor DNA (ctDNA) after resection, and patients with localized GIC (other than PDAC) with persistently elevated ctDNA after resection (GIC). These patients need systemic therapies that can prevent recurrence by eradicating occult micrometastatic disease.

-We have safely treated patients with metastatic GIC using adoptive cell transfer (ACT) autologous tumor-infiltrating lymphocytes (TIL) and with peripheral blood lymphocytes transduced with a T-cell receptor (TCR) specific for a shared hot-spot mutation in KRAS

or TP53 (TCR T-cell therapy). We have demonstrated that TIL can mediate long-term responses in patients with metastatic GIC, providing proof of concept that cell transfer can be effective in low tumor mutational burden, microsatellite stable epithelial cancers, and

can eradicate occult micrometastatic disease. Now, we have also demonstrated that TCR T-cell therapy directed against KRAS G12D, KRAS G12V, and TP53 R175H can mediate objective responses in metastatic GIC.

-Despite some success, practical and theoretical barriers have hampered the translation of TCR T-cell therapy for metastatic GIC. There is evidence that late-stage disease and especially a higher disease burden is associated with resistance to immunotherapy.

Moreover, accumulated toxicity from exposure to cytotoxic chemotherapy may damage the lymphocytes on which TCR T-cell therapy depends. Finally, patients with extensive history of progressive cancer and chemotherapy exposure have depleted physiologic

reserves which can hamper their tolerance of and recovery from cellular therapy. Given these considerations, cellular therapy could be more effective and better tolerated in patients who have a lower burden of disease and are earlier in their disease course.

Objective:

-To determine recurrence-free survival (RFS) (using Response Evaluation Criteria in Solid Tumors [RECIST] v1.1 criteria) of participants treated with TCR T-cells (Arm 1) versus no experimental therapy (Arm 2).

Eligibility:

* Age >= 18 years and <= 72 years.
* PDAC, CRLM, or GIC as follows:

  * PDAC

    * Resected PDAC of stage I-III, and history of detectable ctDNA after resection/local treatment of all known disease.

OR

---If stage I-III, has a history of abnormally elevated cancer antigen (CA)19-9 at diagnosis (before surgery) AND a history of abnormally elevated post-operative CA19-9 after surgery AND a relative increase of post-operative CA19-9 of 2.6-fold compared to the participant s post-operative baseline, as confirmed by two separate tests at least 3 weeks apart.

OR

* Had metastatic disease (stage IV) at diagnosis and were down staged with chemotherapy and underwent resection.

  --CRLM
* Stage IV colorectal cancer with metastases that were completely treated with local therapy and have a history of detectable ctDNA after resection/local treatment of all known disease.

  --GIC
* Participants with resected gastroesophageal cancer, hepatocellular cancer, cholangiocarcinoma, duodenal, small bowel or primary colorectal cancer (i.e., pathologic stage I-III as distinguished from CRLM) and history of detectable ctDNA after resection/local treatment of all known disease.

  * No evidence of measurable disease.
  * History of:

    * KRAS G12D mutation plus HLA-A*11:01
    * KRAS G12D mutation plus HLA-C*08:02
    * KRAS G12V mutation plus HLA-C*01:02
    * TP53 R175H mutation plus HLA-A*02:01
  * Adequate basic laboratory values

Design:

* Eligible participants will be randomized in a 1:1 fashion after successful completion of apheresis under 03-C-0277 and verification of a sufficient PBL sample for use for TCR Tcell therapy.
* Participants randomized to Arm 1 will return to NIH to receive TCR T-cells plus aldesleukin following lymphodepletion with reduced-dose cyclophosphamide and fludarabine. Participants randomized to Arm 2 will return to the NIH for surveillance.
* There will be three strata for randomization:

  1. Pancreas cancer
  2. Stage IV colorectal cancer
  3. Other gastrointestinal cancers (including stage I-III colorectal cancer)
* TCR T-cells are generated by transduction of autologous peripheral blood lymphocytes (PBL) with TCR genes encoding a T-cell receptor that recognizes a hotspot mutation in KRAS G12D, KRAS G12V, or TP53 R175H in the context of HLA.
* Participants randomized to Arm 2 will receive no experimental therapy but will have serial clinical evaluation and surveillance on the same schedule as participants in Arm 1.
* Baseline clinical evaluation and radiographic assessment will be performed on all participants before randomization, and both arms will undergo radiographic evaluation on the same schedule every 3-6 months thereafter.
* It is anticipated that approximately two participants per month will be randomized. There will be a limit of 30 evaluable participants per Arm for a total of 60 evaluable participants. Thus, the accrual may be completed in approximately 2.5 years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Resected pancreas ductal adenocarcinoma (PDAC):

  * Resected pancreas ductal adenocarcinoma
  * If stage I-III has a history of detectable circulating tumor DNA (ctDNA) after resection/local treatment of all known disease.

OR

--If stage I-III, have a history of abnormally elevated cancer antigen (CA)19-9 at diagnosis (before surgery) AND a history of abnormally elevated post-operative CA19-9 measured at least 30 days after surgery AND a history of the relative increase of postoperative CA19-9 of 2.6-fold or more compared to the participant s post-operative baseline, as confirmed by two separate tests at least 3 weeks apart.

OR

* Had metastatic disease (stage IV) at diagnosis and were down staged with chemotherapy and underwent resection.

  -Colorectal liver, lung, and/or lymph node metastases (CRLM):
* Participants with stage IV colorectal cancer with metastases to the liver, lung, and/or lymph nodes that were completely treated with local therapy (resection, ablation, and/or radiotherapy).
* Must have a history of detectable ctDNA after resection/local treatment of all known disease.

  -Gastrointestinal carcinoma (GIC):
* Participants with resected gastroesophageal cancer, hepatocellular cancer, cholangiocarcinoma, duodenal, small bowel, or primary colorectal cancer (i.e., pathologic stage I-III as distinguished from CRLM).
* Must have a history of detectable ctDNA after resection/local treatment of all known disease.

  * Confirmation of diagnosis of cancer by the NCI Laboratory of Pathology (LP).
  * Must have a history of:
* KRAS G12D mutation plus HLA-A*11:01

OR

--KRAS G12D mutation plus HLA-C*08:02

OR

--KRAS G12V mutation plus HLA-C*01:02

OR

* TP53 R175H mutation plus HLA-A*02:01.

  -Treated with standard systemic and/or radiotherapy if indicated unless participant refusal or non-tolerance of the standard regimen. For example:
* Participants with PDAC should receive neoadjuvant or adjuvant chemotherapy (5-FU or gemcitabine-based).
* Participants with CRLM should have received at least one line of 5FU-based chemotherapy (i.e., FOLFOX or FOLFIRI).
* Participants with resected stage III colon cancer should have received 5FU-based adjuvant therapy (i.e., FOLFOX or FOLFIRI).

  * CRLM only: Participants with a history of brain metastases that have been treated with stereotactic radiosurgery or resection must be clinically stable for 3 months after treatment to be eligible.
  * Age >= 18 years and <= 72 years.
  * Clinical performance status of ECOG 0 or 1
  * Individuals of child-bearing potential (IOCBP) must agree to use highly effective contraception (hormonal, intrauterine device [IUD], abstinence, surgical sterilization) at the study entry and up to and 12 months after the last dose of combined chemotherapy. Individuals that can father children must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) at the study entry and up to 4 months after the last dose of study drugs. We also will recommend individuals that can father children with partners that can bear children ask their partners to be on highly effective birth control (hormonal, IUD, surgical sterilization). Individuals that can father

children must not freeze or donate sperm within the same period.

NOTE: IOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.

* Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 4 months after the last dose of the study drug(s).
* Viral testing

  * Seronegative for human immunodeficiency virus (HIV) antibody.
  * Negative for hepatitis B (HBV) surface antigen (HbsAg), and seronegative for hepatitis C (HCV) antibody. If the HCV antibody test is positive, then the participant must be tested for the presence of antigen by RT-PCR and be HCV RNA negative to be eligible.
* Hematology

  * Absolute neutrophil count (ANC) > 1000/mm^3 without the support of filgrastim
  * White blood cells (WBC) >= 2500/mm^3
  * Platelet count >= 80,000/mm^3
  * Hemoglobin > 8.0 g/dL.
* Chemistry

  * Alanine aminotransferase (ALT) <= 5.0 x upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) <= 5.0 x ULN
  * Creatinine <= 1.6 mg/dL
  * Total bilirubin <= 2.0 mg/dL, except in participants with Gilbert s Syndrome, who must have a total bilirubin < 3.0 mg/dL.
* Four weeks must have passed after any prior systemic therapy for cancer, any investigational agents, surgical procedures, or limited field radiotherapy prior to randomization, as long as related major organ toxicities have recovered to grade 1 or less per Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.

NOTE: Participants with adverse events Grade 2 that are deemed irreversible and stable and will not prevent administration of the study drug(s)/intervention or prevent compliance with the study requirements (e.g., alopecia, peripheral neuropathy, laboratory parameters not

otherwise specified per the eligibility criteria) are an exception to this criterion and are eligible.

* Ability of the participant to understand and the willingness to sign a written informed consent document.
* Willing to sign a durable power of attorney.
* Participants must be co-enrolled on protocols 03-C-0277 (Cell Harvest and Preparation for Surgery Branch Adoptive Cell Therapy Protocols), and 09-C-0161 (Follow-up Protocol for Subjects Previously Enrolled on NCI Surgery Branch Studies).

EXCLUSION CRITERIA:

* Unequivocal radiographic evidence of residual tumor.
* Participants with measurable disease per RECIST v1.1 criteria.
* Any form of secondary immunosuppression.
* Active or chronic infections requiring anti-microbial, anti-fungal, or anti-viral treatment.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and Acquired immunodeficiency syndrome [AIDS]).
* History of major organ autoimmune disease.
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or aldesleukin.
* History of coronary revascularization or ischemic symptoms.
* Left ventricular ejection fraction (LVEF) <= 45% for participants with a clinical history prompting cardiac evaluation (e.g., participants who are >= 65 years of age, or who have a history of ischemic heart disease, chest pain, or clinically significant atrial and/or ventricular arrhythmias, including but not limited to atrial fibrillation, ventricular tachycardia, heart block OR Participants < 65 years of age with cardiac risk factors [e.g., diabetes, hypertension, obesity]).
* Forced expiratory volume in the first second (FEV1) <= 50% predicted for participants with a clinical history prompting pulmonary evaluation (e.g., a prolonged history of cigarette smoking [>= 20 pack-year smoking history within the past two years], symptoms

of respiratory dysfunction, thoracic surgeries, or other clinical indications).

* Positive beta-human chorionic gonadotropin (beta-HCG) serum or urine pregnancy test performed in IOCBP at screening.
* Uncontrolled intercurrent illness evaluated by medical history and physical exam that are not stable and would potentially increase the risk to the participant.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-09 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) | 12 weeks then every 3 months x 3, every 6 months after that until progression or 5 years since randomization.
  RFS will be assessed with tumor markers and radiographic findings in each group and reported using the Kaplan-Meier method with 95% confidence intervals on the median RFS in each group.

SECONDARY OUTCOMES:
Overall survival (OS) | 12 weeks then every 3 months x 3, every 6 months after that until progression or 5 years since randomization. After progression contact with participants every 6 months until the first of death or 5 years after randomization.
  OS will be assessed in each group and reported using the Kaplan-Meier method with 95% confidence intervals on the median OS in each group.
Safety | until 6 months after the last dose of study agents
  The number and frequency of adverse events for group 1 participants as assessed per CTCAE version 5. Safety will be analyzed by reporting the number of patients experiencing toxicity, classified by type and grade to the experimental regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas D Klemen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared after reaching the primary endpoint per the identified timeframe.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001870-C.html